CLINICAL TRIAL: NCT03945630
Title: Quadratus Lumborum Block in Total Hip Arthroplasty - Effect on Analgesia and Early Physiotherapy: a Randomised Controlled Trial
Brief Title: Quadratus Lumborum Block in Total Hip Arthroplasty - Effect on Analgesia and Early Physiotherapy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit patients due to COVID19
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Radoslaw Owczuk, Professor, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MK-1
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Total Hip Arthroplasty
Keywords: Quadratus Lumborum Block
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: * Procedure: Quadratus Lumborum Block (QLB) Ultrasound guided Quadratus Lumborum block using an anterior approach. (QLB3; TQL-Transmuscular Quadratus Lumborum)
  * Procedure: Standard of Care (no QLB)
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- anterior Quadratus Lumborum Block (QLB) (Experimental): Anterior QLB will be performed in the sitting position. This block is also known as TQL- Transmuscular QLB or QLB 3. A convex transducer will be placed in a transverse position, in the posterior axillary line and tilted caudad until the 'shamrock sign' at L4 level will be obtained. An 80-110 mm SonoTAP (PAJUNK Medizintechnologie, Geisingen, Germany) will be inserted in-plane from the lateral end of the transducer and advanced until the needle tip will be inside the interfascial plane between the Quadratus Lumborum and the Psoas muscles. The successful needle placement will be confirmed by observing the spread of 5 mls 0,9%NaCl. Subsequently, 30 ml 0.5% ropivacaine with 100 mcg dexmedetomidine and adrenaline 1:200,000 will be injected. Satisfactory interfascial spread will be assessed by longitudinal probe orientation.
  Following QLB, a spinal anaesthetic will be sited and a THA via posterior approach will be performed.
  Interventions: Procedure: anterior Quadratus Lumborum Block
- Standard of Care (no QLB) (Active Comparator): A spinal anaesthetic will be sited and a THA via posterior approach will be performed.
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Procedure: anterior Quadratus Lumborum Block — Interfascial plane block
  Other Names: TQL; Transmuscular QLB; QLB 3
  Arms: anterior Quadratus Lumborum Block (QLB)
Procedure: Standard of Care — No QLB
  Arms: Standard of Care (no QLB)

SUMMARY:
Currently there is no consensus on the optimal peripheral nerve block for Total Hip Arthroplasty (THA). Furthermore, there is a gap in the literature in regard to the efficacy of Quadratus Lumborum Block (QLB) for Total Hip Arthroplasty via posterior approach.

This Randomised Controlled Trial aims to examine the effectiveness of anterior QLB in patients undergoing Total Hip Arthroplasty via posterior approach. The investigators hypothesise that anterior QLB and spinal anaesthesia is superior to spinal anaesthesia alone with reference to analgesic efficacy and functional ability to engage with physiotherapy in the first 24 hours postoperatively.

DETAILED DESCRIPTION:
Adequate analgesic strategies for Total Hip Arthroplasty (THA) are of paramount importance in early rehabilitation and enhanced recovery. Ultrasound guided peripheral nerve blocks emerge as the key element of multi-modal analgesia in modern orthopaedic surgery, but in this setting, given the complex sensory innervation of the hip joint, the optimal regional technique for THA is yet to be elucidated. Many centres incorporate Suprainguinal Fascia Iliaca Block in their THA regimen. Although it confers certain benefits, its analgesic efficacy may be suboptimal for posterior approach THA, especially with regards to dermatomal sensory distribution. The Quadratus Lumborum Block (QLB) is a relatively novel technique, yet its role is already established in providing somatic and visceral analgesia for abdominal and pelvic surgery. There are case reports indicating its utility in THA; Adhikary et al. report that QLB is non inferior to Lumbar Plexus Block in terms of its analgesic efficacy, while being easier to perform and carrying less risks.

There remains some debate regarding the QLB mechanism of action. Its clinical effect may be attributed to the spread to thoracic and lumbar paravertebral spaces, spread within the thoracolumbar fascia or even direct spread to the lumbar plexus branches; perhaps all three mechanisms are involved. Thus, QLB is biologically plausible to provide analgesia without significant motor block for posterior approach THA, but for that purpose, neither the optimal volume of local anaesthetic nor the site of injection (anterior vs posterior vs lateral QLB or the vertical height of injection endpoint) have been established in the literature. Based on the available evidence, as well as experience at our institution, the investigators hypothesise, that in patients undergoing THA via posterior approach, anterior QLB at L4 level using 30 ml 0,5% ropivacaine, 100mcg dexmedetomidine and 1:200,000 adrenaline will reduce movement pain scores within the first 24hours, without clinically significant motor block.

The participants will be randomised into one of two groups using an internet based randomisation tool (https://www.randomizer.org/), and subsequently allocated to either group, with the allocation concealed in a sealed opaque envelope.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral total hip arthroplasty
* Adults 18 - 90 years.
* ASA classification of I, II or III

Exclusion Criteria:

* Patients with allergies to local anaesthetic
* Patients with pre-existing neurologic or anatomic deficits in the lower extremity on the side of the operation
* BMI > 40
* Extremes of stature (145cm > Height >210cm)
* Patients with co-existing coagulopathy
* Patients refusing spinal anaesthetic or regional block
* Revision hip arthroplasty
* Contraindications to spinal anaesthetic
* Unsatisfactory confirmation of the local anaesthetic spread in the interfascial plane
* Patients requiring transfusion > 2 units of Red Packed Cells in the postoperative period

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
NRS score during mobility assessment with physiotherapist | 24 hours
  Postoperative movement pain score using an 11-point Numeric Rating Scale (NRS) (0- no pain; 10- the worst pain imaginable) during the first postoperative mobility assessment by physiotherapist

SECONDARY OUTCOMES:
Serial postoperative NRS pain scores (rest and movement) | Time Frame: 3 hours after intervention. 6 hours after intervention. At 22:00 hour on Day 0. At 6:00 hour on Day 1. 36 hours after intervention
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain (0- no pain; 10- the worst pain imaginable). The investigators will record pain score at rest at the specified time intervals; except at 6 hours after intervention (block sited), when the pain score will be recorded simultaneously with hip range of motion assessment
Opioid consumption | 48 hours
  Opioid consumption (oxycodone)
Time to first request for rescue opioid analgesia | 48 hours
  Time to first request for a rescue opioid administration (PRN oxycodone)
Ability to ambulate with physiotherapist | up to 24 hours
  Distance in metres will be recorded during the first attempt to ambulate with physiotherapist (usually on Day 1)
Operated limb sensory block | 6 hours after intervention. Within 24 hours (during the first attempt to ambulate with physiotherapist)
  The level of sensory block (to cold temperature), tested with cold spray, will be recorded by a trained assessor on the dermatome map chart.
Operated limb muscle weakness | 6 hours after intervention. Within 24 hours (during the first attempt to ambulate with physiotherapist)
  QLB's effect on muscles involved in hip joint movement will be evaluated. Additionally, muscles innervated by major motor nerves originating in the Lumbar and Sacral plexuses will be examined. The investigators will test patient's ability to perform the motor tasks below, using a 6-point Oxford scale (0 represents no muscle movement and 5 corresponds to normal strength):
  hip abduction, straight leg raise, heel slide, knee extension (while supporting the knee under the popliteal fossa), foot plantar flexion, foot dorsal flexion.
Total operation time | During the expected duration of anaesthesia and surgery, which is on average 3 hours
  Start to end of the recorded anaesthesia time (that includes the operation time)
Length of Stay in Recovery area | Expected 30 minutes to 3 hours
  Length of Stay in Recovery area in minutes
The incidence of nausea and/or vomiting | 48 hours
  The incidence of nausea and/or vomiting (the total number recorded)
Patient satisfaction with anaesthesia | up to 6 days
  Patient satisfaction with anaesthesia data will be collected on discharge from hospital on a scale of 0-4 (0=very dissatisfied, 4= very satisfied)
Overall patient satisfaction | up to 6 days
  Overall patient satisfaction data will be collected on discharge from hospital on a scale of 0-4 (0=very dissatisfied, 4= very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Kaminski, Principal Investigator — Medical University of Gdańsk, University Clinical Centre, Gdansk
Locations (1):
- Medical University of Gdańsk - Departament of Anesthesiology and Intensive Care, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided